CLINICAL TRIAL: NCT00644696
Title: A Phase One Study of Intravenous Irinotecan and Bortezomib in Children With Recurrent/Refractory High-Risk Neuroblastoma
Brief Title: Study of Irinotecan and Bortezomib in Children With Recurrent/Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.084; HUM 7859 (Other: University of Michigan Medical School IRB)
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Irinotecan; Bortezomib
MeSH Terms: conditions — Neuroblastoma | interventions — Irinotecan; Bortezomib; Cefpodoxime; Cefixime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan and Bortezomib (Experimental): Irinotecan and Bortezomib will both be administered
  Interventions: Drug: Irinotecan and Bortezomib

INTERVENTIONS:
Drug: Irinotecan and Bortezomib — Dose level-1a: IV Irinotecan 30 mg/m2/day, IV bortezomib 1.2mg/m2/day Dose level-1: IV Irinotecan 35 mg/m2/day, IV bortezomib 1.2mg/m2/day Dose level-2: IV Irinotecan 40 mg/m2/day, IV bortezomib 1.2mg/m2/day Dose level-3: IV Irinotecan 45 mg/m2/day, IV bortezomib 1.2mg/m2/day Dose level-4: IV Irinotecan 50 mg/m2/day, IV bortezomib 1.2mg/m2/day
  Other Names: Velcade; Cefpodoxime; Cefixime

SUMMARY:
This Phase One pediatric trial seeks to take advantage of the susceptibility of neuroblastoma to proteasome inhibitors, proven in vitro, along with the proven in vitro synergy of bortezomib with irinotecan and the successful Phase One pediatric trials of bortezomib to create a treatment using these two drugs in combination to treat refractory/recurrent neuroblastoma in children and young adults 25 and under.

DETAILED DESCRIPTION:
In spite of intensive treatment including high-dose chemotherapy with autologous peripheral stem cell transplantation and radiation therapy, the long-term survival of patients with high-risk neuroblastoma remains poor. Patients who experience a relapse of their disease or fail to achieve complete remission fare even worse. More intense chemotherapy is not the answer. The development of new drugs with different mechanisms of action are required.

Inhibitors of the proteasome have created a considerable interest in their use in cancer chemotherapy, either as a single agent or in combination with other chemotherapeutic agents. The precise mechanism of action for these class of drugs is unclear, however, inhibition of I-kB degradation by VELCADE® (bortezomib) decreases NF-kB activity in neuroblastoma cell lines as well as other systems.

Previous studies have reported the activity of Irinotecan, a strong Topoisomerase-I inhibitor, against murine xenografts including those with high-risk features such as MYCN gene amplification (MYCN is also called V-Myc Myelocytomatosis Viral Related Oncogene, Neuroblastoma Derived). Irinotecan has also been shown to be active against neuroblastoma xenografts resistant to vincristine, melphalan, and topotecan, suggesting an alternative mechanism of resistance to Irinotecan. In vitro synergy between bortezomib and irinotecan has been documented in pancreatic cancer by others and in neuroblastoma by our group.

ELIGIBILITY:
Inclusion Criteria:

* No greater than 25 years of age when originally diagnosed.
* Histologic verification of condition.
* Has recurrent/progressive; or resistant/refractory neuroblastoma with at least ONE of the following:

  1. Measurable tumor on MRI or CT scan or X-ray (at least 20 mm in at least one dimension) or
  2. MIBG scan with positive uptake at minimum of one site, or
  3. Bone marrow with tumor cells seen on routine morphology (not by NSE staining only) of bilateral aspirate and/or biopsy on one bone marrow sample.
* Has Lansky or Karnofsky score of 60%, and a life expectancy of > 2 months.
* Has fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy.
* Has not received treatment with myelosuppressive agents within 3 weeks and with any biological therapy within 2 weeks of study entry.
* Has not received radiation for a minimum of four weeks prior to study entry at the site of any lesion that was biopsied to document study eligibility.
* Patient is 2 months post myeloablative therapy and autologous stem cell transplant.
* At least six weeks must have elapsed since treatment with therapeutic doses of MIBG.
* Patients who have previously received combination bortezomib and irinotecan are ineligible but can have received one of the drugs.
* Must not have received hematopoietic growth factors within 2 days of study entry.
* Cannot be receiving enzyme-inducing anticonvulsants (phenobarbital, phenytoin, carbamazepine).
* Concomitant radiotherapy to painful bone lesions will be allowed (excluding intestinal tract, spine or pelvis) but other non-radiated sites of measurable disease must be available to assess response to chemotherapy.
* Patient has adequate bone marrow function (defined).
* Patient has adequate renal function (defined).
* Patient has adequate liver function (defined).
* Post-menarchal females must have a negative pregnancy test measuring beta-human chorionic gonadotropin(HCG). All males and females must use effective contraception during study.

Exclusion Criteria:

* Patient is status post-allogenic stem cell transplant.
* Patient has uncontrolled infection or active diarrhea defined as 2 or more stools per day greater than baseline.
* Presence of HIV, active hepatitis B, or active hepatitis C infection.
* Pregnancy, as determined by Beta-human chorionic gonadotropin(HCG)measurement.
* Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or various other indications of heart disease. (defined)
* Hypersensitivity to bortezomib, irinotecan, cefixime, boron or mannitol.
* Female subject is breast-feeding.
* Serious medical or psychiatric illness likely to interfere with participation.
* Patient has received other investigational drugs within 14 days before enrollment.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determine highest dose of IV irinotecan administered in conjunction with bortezomib without causing severe side effects. | 3 years

SECONDARY OUTCOMES:
Measure the neuroblastoma tumors after treatment with irinotecan and bortezomib to determine whether there was a change in size. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajen Mody, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States